CLINICAL TRIAL: NCT04296422
Title: Evaluation of the Effect of Different Acupuncture Dose on Premenstrual Syndrome and the Relationship Between Premenstrual Syndrome and TCM Syndrome Complex
Brief Title: Different Does of Acupuncture on Premenstrual Syndrome Efficacy Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-10712111
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Premenstrual Syndrome
Keywords: Acupuncture; Premenstrual Syndrome; TCM syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Anti-Inflammatory Agents, Non-Steroidal; Naproxen; Diclofenac; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Gynecologic Treatment group (Active Comparator): Taking NSAIDs or oral contraceptives.NSAIDs include Ibuprofen, Naproxen, Diclofenac, and Piroxicam. Oral contraceptives include Yasmin.
  Interventions: Drug: NSAIDs or oral contraceptives treatment
- Low dose acupuncture group (Experimental): Acupuncture has fewer acupuncture points.
  Interventions: Device: Low dose acupuncture
- High dose acupuncture group (Experimental): Acupuncture has more acupuncture points.
  Interventions: Device: High dose acupuncture

INTERVENTIONS:
Drug: NSAIDs or oral contraceptives treatment — Taking NSAIDs or oral contraceptives.NSAIDs include Ibuprofen, Naproxen, Diclofenac, and Piroxicam. Oral contraceptives include Yasmin.
  Other Names: Taking NSAIDs or oral contraceptives.NSAIDs include Ibuprofen, Naproxen, Diclofenac, and Piroxicam. Oral contraceptives include Yasmin.
  Arms: Conventional Gynecologic Treatment group
Device: Low dose acupuncture — Six acupoints: Three Yin Intersection( SP6)、Grandfather Grandson(SP4)、 Sea of Blood(SP10) 、Sea of Qi(RN6)、Origin Pass(RN4) 、Inner Pass(PC6)
  Arms: Low dose acupuncture group
Device: High dose acupuncture — Twelve acupoints: Three Yin Intersection( SP6)、Grandfather Grandson(SP4)、 Sea of Blood(SP10) 、Sea of Qi(RN6)、Origin Pass(RN4) 、Middle Extremity(RN3)、Inner
  Arms: High dose acupuncture group

SUMMARY:
The design of the study includes 3 groups for women with premenstrual syndrome, 1low dose acupuncture in the low-dose group, 2 high dose acupuncture in the high-dose group, and 3 the drug group (contraceptives) . Serum marker change of PGE2, CA125, E2, and progesterone in enrolled patients will be measured before and after treatment, along with VAS and MDQ questionnaires. The treatment efficacy of different groups and the relationship between PMS and patients TCM syndrome pattern will also be recorded and estimated.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is the sum of a group of symptoms (including physical and psychological symptoms) that occurs during the luteal phase of the menstrual cycle. Women who have such symptoms have been estimated as high as 75%; of which 3% to 8% are severe symptoms, called premenstrual dysphoric disorder (premenstrualdysphoric syndrome, PMDD). The two groups are very similar. PMS is mostly for physical discomfort, while PMDD is for emotional problems, affecting women's sleep seriously.

Regarding the treatment of premenstrual syndrome (PMS), western medicine adopt oral contraceptive pills (OCP) as the first-line medication. However, the common side effects of OCP, such as headache, dizziness, nausea, vomiting, depression, breast pain and so on are also troublesome, In recent years, some women also use acupuncture as an adjunctive replacement therapy because of its safety and fewer side effects. Nevertheless, the factors affecting treatment effect of acupuncture and moxibustion. such as the selection of acupoint s ( of which meridians) or number(dose) of acupuncture ,etc., maight affect the efficacy, yet the relevant research on this issue is not enough. In traditional Chinese medicine theory, acupuncture and moxibustion regulate the energy of the meridians and adjust blood and qi, which in turn help the balance of yin and yang. Female menstrual cycle is a process of conversion between yin and yang in TCM theory. While in western medicine, it is regulated by the endocrine system.

ELIGIBILITY:
Inclusion Criteria:

1.15 to 49 years 2.with a history of regular menstrual cycles (28days±7 days) 3.Symptoms：breast pain、dizziness、bloating、cramps、nausea、vomiting、 diarrhea、headache、 fatigue，etc

Exclusion Criteria:

1. irregular menstrual cycles
2. intrauterine contraceptive device (IUCD/IUD)
3. uncontrolled neurological diseases
4. lactation， pregnant women，or those with plans to get pregnant in the coming half year

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-18 (Estimated); Study Completion 2020-09-18 (Estimated)

PRIMARY OUTCOMES:
Wang Qi Chinese Medicine Questionnaire | Change from Baseline TCM constitutions at 4 cycles (each cycle is 30 days).
  This questionnaire is used to survey TCM constitutions. Evaluate body constitution of

SECONDARY OUTCOMES:
Visual analogue scale(VAS) score | Change from Baseline VAS score at 4 cycles (each cycle is 30 days).
  VAS is used to assess the extent of menstrual pain.
Blood test estrogen | Change from Baseline blood test at 4 cycles (each cycle is 30 days).
Blood test progesterone | Change from Baseline blood test at 4 cycles (each cycle is 30 days).
Blood test prostaglandin | Change from Baseline blood test at 4 cycles (each cycle is 30 days).
Menstrual Distress Questionnaire(MDQ) | Change from Baseline Menstrual Distress Questionnaire at 4 cycles (each cycle is 30 days).
  Contain: Pain；Concentration；Behavioral Change；Autonomic Reactions；Water Retention；Negative Affect

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Ju Chien, Principal Investigator — Taipei City Hospital; Yi-Shuo Huang, Study Director — Taipei City Hospital
Locations (1):
- Taipei City H, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study will have a continuous plan.